CLINICAL TRIAL: NCT00422591
Title: Prospective Evaluation of Standard Chemotherapy Regimen of Idarubicin and Cytarabine in Patients With Newly Diagnosed Acute Myeloid Leukemia (AML)
Brief Title: Standard Idarubicin and Cytarabine for the Treatment of Acute Myeloid Leukemia (AML)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-0813; NCI-2012-01412 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2007-01-16; First posted 2007-01-17 (Estimated); Results first posted 2018-06-12 (Actual); Last update posted 2018-08-23 (Actual); Status verified 2018-07

CONDITIONS: Leukemia; Acute Myeloid Leukemia; AML
Keywords: Cytarabine, Idarubicin; Leukemia; Acute Myeloid Leukemia; AML; Cytarabine; Idarubicin
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute | interventions — Cytarabine; Idarubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Idarubicin + Cytarabine (Experimental): Idarubicin 12 mg/m2 IV over 1 hour daily x 3 (days 1-3). Cytarabine 1.5 g/m2 IV over 24 hours daily on day 1-4 (age <60 years) or days 1-3 (age > 60 years).
  Interventions: Drug: Cytarabine; Drug: Idarubicin

INTERVENTIONS:
Drug: Cytarabine — 1.5 g/m2 IV over 24 hours daily on day 1-4 (age <60 years) or days 1-3 (age > 60 years).
  Other Names: Ara-C; Cytosar-U
Drug: Idarubicin — 12 mg/m2 IV over 1 hour daily x 3 (days 1-3)
  Other Names: Idamycin®

SUMMARY:
The goal of this clinical research study is to find out if standard chemotherapy given with idarubicin and Cytarabine (ara-C) can help to control AML.

Objectives:

To determine the complete response (CR) rate, event-free survival (EFS) and overall survival (OS) of patients with newly diagnosed acute myeloid leukemia (AML) receiving standard combination chemotherapy with Idarubicin and cytarabine.

DETAILED DESCRIPTION:
Ara-C and idarubicin are designed to interfere with DNA's (the genetic material of cells) ability to repair itself, causing cancer cells to die.

If you are found to be eligible to take part in this study, you will receive treatment with idarubicin and ara-C for up to 8 cycles. One cycle lasts about 4-5 weeks. Cycles 1 and 2 are called induction therapy, which is used to help induce (cause) a remission. Cycles 3 to 8 are called consolidation therapy, which is a type of high-dose chemotherapy often given as the second phase of a cancer treatment.

After Cycle 1, you will have a brief rest period of a few days, before you move on to Cycle 2. On Day 1 of Cycle 1, you will receive cytarabine by vein as a continuous infusion over 4 days. It will only be 3 days if you are age 60 or older. On Days 1-3 of Cycle 1, you will receive idarubicin by vein over 1 hour once a day.

The dose of the study drugs you receive may be changed to help manage side effects (such as nausea and diarrhea) that you may experience. Medications (given by mouth or by vein), such as Tylenol (acetaminophen), may be given before and during treatment to help decrease the risk of such side effects. The study doctor will specify what these medications are.

You will have blood drawn (about 2 teaspoons) for routine tests about once a week during treatment. Starting on Days 21-28, you will have bone marrow collected every 1-2 weeks to check the status of the disease. Blood (about 2 tablespoons) will also be drawn at least twice a week after each cycle of therapy (beginning about 4-6 weeks from the start of treatment each cycle) to check your blood counts.

Cycle 2 will begin after your blood counts have recovered. If at the end of Cycle 1 you have not achieved a remission (disease has decreased), you may receive Cycle 2, which will be similar to Cycle 1.

If the disease is responding to treatment after Cycle 2 (after completion of induction therapy), you will receive up to 6 more cycles of therapy. These cycles are called consolidation therapy. Consolidation therapy is a type of high-dose chemotherapy often given as the second phase to treat cancer. For consolidation therapy, you will receive ara-C as a continuous infusion over 3 days starting on Day 1 of Cycle 3. On Days 1 and 2 of Cycles 3 and 4, you will receive idarubicin by vein over 1 hour. Your blood (about 2 tablespoons) will be drawn at least twice a week after each cycle to check your blood counts. Cycle 3 will begin after your blood counts have recovered.

After completion of consolidation therapy, you may receive what is called maintenance therapy. Maintenance therapy will start after completion of consolidation therapy. Maintenance therapy is often given to help keep cancer in remission. It is treatment that is given to help the original treatment keep working. You will be told if you will have maintenance therapy as well as the drugs and drug schedule you will be on.

During consolidation and/or maintenance therapy, blood (about 2 teaspoons) will be drawn for routine tests every 1-2 weeks. You will have bone marrow collected every 3-6 months to check the status of the disease.

You may have treatment on this study for up to 8 cycles (induction and consolidation therapy) or more (for maintenance therapy), depending on disease response to the study drugs. If the disease gets worse or you experience any intolerable side effects, you will be taken off this study, and your study doctor will discuss other treatment options with you.

Once your participation is over on this study, you will be followed-up with a phone call by the study doctor or study nurse to check on how you are doing and if you have experienced any intolerable side effects. The call should last about 10-15 minutes.

This is an investigational study. Idarubicin and ara-C are both FDA approved and commercially available. Up to 200 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of 1) AML (WHO classification definition of >/= 20% blasts). Patients with M6 AML with less than 20% blasts are eligible.
2. Patients aged 15 to 75 years are eligible. Patients must be chemo-naïve, i.e. not have received any prior chemotherapy (except hydrea) for AML. They could have received transfusions, hematopoietic growth factors or vitamins. Temporary measures such as pheresis or hydrea (0.5 to 5g daily or more for up to 3 days) are allowed .
3. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0, 1, 2, or 3 at screening.
4. Serum biochemical values with the following limits: - creatinine </= 2.0 mg/dl - total bilirubin </= 2.0 mg/dL, unless increase is due to hemolysis - transaminases (SG PT) </= 3x upper limit of normal (ULN)
5. Ability to understand and provide signed informed consent.

Exclusion Criteria:

1. Subjects with Acute Promyelocytic Leukemia (APL).
2. Presence of active systemic infection.
3. Any coexisting medical condition that in the judgment of the treating physician is likely to interfere with study procedures or results.
4. Nursing women, women of childbearing potential with positive urine pregnancy test, or women of childbearing potential who are not willing to maintain adequate contraception (such as birth control pills, intrauterine device (IUD), diaphragm, abstinence, or condoms by their partner) over the entire course of the study.

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2006-12; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Farhad Ravandi-Kashani, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 12/2006 to 01/2017
Pre-assignment Details: Of the 175 participants registered, six were never treated.
Groups:
- Idarubicin + Cytarabine: Idarubicin 12 mg/m2 intravenously (IV) over 1 hour daily days 1-3. Cytarabine 1.5 g/m2 IV over 24 hours daily on day 1-4 (age <60 years) or days 1-3 (age > 60 years).
Period: Overall Study
Arm/Group | Idarubicin + Cytarabine
Started | 175
Completed | 169
Not Completed | 6
Not completed — Physician Decision | 4
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Idarubicin + Cytarabine
Number analyzed (Participants) | 175
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 156
  >=65 years | 19
Age, Continuous [Median (Full Range); unit: years] | 55 [19 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77
  Male | 98
Region of Enrollment [Number; unit: participants]
  United States | 175

OUTCOME MEASURES:

1. Primary Outcome: Complete Response (CR) Rate
Description: Complete Response (CR): Normalization of marrow (< 5% blasts; >10% cellularity) and of peripheral blood counts (no circulating blasts, neutrophil count > 109/L, platelet count > 100 x 109/L).
Time Frame: Up to 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Idarubicin + Cytarabine
Number analyzed (Participants) | 169
Participants
  Complete Response | 98
  Partial Response | 4
  Complete Response w/o Platelet Recovery | 9
  Death | 7
  No Response | 51

2. Secondary Outcome: Event-Free Survival (EFS)
Description: Event -Free Survival (EFS) EFS was calculated with Kaplan-Meier estimates. Event-free survival (EFS), defined as the time to no response to intensive induction therapy, relapse, or death of any cause, whichever comes first.
Time Frame: from treatment initiation until treatment failure, relapse, or death
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Idarubicin + Cytarabine
Number analyzed (Participants) | 169
Months | 4.7 [1 to 72]

3. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival (OS) was calculated with Kaplan-Meier estimates. OS was calculated from the time of treatment initiation until death.
Time Frame: Until death or loss of follow-up
Measure: Median (Full Range); unit: Months
Arm/Group | Idarubicin + Cytarabine
Number analyzed (Participants) | 169
Months | 11.3 [1 to 75]

ADVERSE EVENTS:
Time Frame: Adverse events captured from the time of participant consent and will be followed to resolution or stabilization; up to 1 year.
Arm/Group | Idarubicin + Cytarabine
All-Cause Mortality (participants affected / at risk) | 10/169
Serious Adverse Events (participants affected / at risk) | 77/169
Other Adverse Events (participants affected / at risk) | 87/169
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Idarubicin + Cytarabine (N=169)
Abscess Left Groin (Skin and subcutaneous tissue disorders) | 1 (1)
Abdominal Pain (General disorders) | 3 (3)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Arrythmia (Cardiac disorders) | 1 (1)
Arthritis Knee (Musculoskeletal and connective tissue disorders) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 2 (2)
Cardiac Arrest (Cardiac disorders) | 1 (1)
Cardiac Infarction (Cardiac disorders) | 1 (1)
Catheter Related Infection (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 2 (2)
Cholecyctectomy (Surgical and medical procedures) | 1 (1)
Cholecystitis (Infections and infestations) | 2 (3)
Clostridium Difficile Colitis (Infections and infestations) | 1 (1)
Colitis (Infections and infestations) | 1 (1)
Death (General disorders) | 10 (10)
Diarrhea (Gastrointestinal disorders) | 4 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Edema - leg (Blood and lymphatic system disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Fever (General disorders) | 6 (7)
Hemorrhage Gastrointestinal (Blood and lymphatic system disorders) | 1 (1)
Hyperbilirubinemia (Blood and lymphatic system disorders) | 1 (1)
Hypotension (Cardiac disorders) | 1 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Infection (Infections and infestations) | 14 (18)
Infection Abcess (Infections and infestations) | 1 (1)
Intracerebral Hemorrhage (Blood and lymphatic system disorders) | 1 (1)
Lung Injury (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Myelosupression (Immune system disorders) | 2 (2)
Neuropathy (Nervous system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Neutropenic Fever (Infections and infestations) | 27 (34)
Pain Cardiovascular (Cardiac disorders) | 1 (1)
Pain Head/Neck (General disorders) | 1 (1)
Pancreatitis (Hepatobiliary disorders) | 1 (1)
Pneumonia (Infections and infestations) | 9 (10)
Pneumonitis (Infections and infestations) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Renal Failure (Renal and urinary disorders) | 2 (2)
Seizure (Nervous system disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Sinus Bradycarida (Cardiac disorders) | 1 (1)
Supraventricular arrhythmia (Cardiac disorders) | 1 (1)
Syncope (Nervous system disorders) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Ventricular Arrhythmia (Cardiac disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Wound Infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Idarubicin + Cytarabine (N=169)
Rash (Skin and subcutaneous tissue disorders) | 20 (20)
Diarrhea (Gastrointestinal disorders) | 26 (26)
Nausea (Gastrointestinal disorders) | 10 (12)
Febrile Neutropenia (Infections and infestations) | 47 (65)
Infection/unknown ANC (Infections and infestations) | 20 (28)
Infection other (Infections and infestations) | 10 (10)
Opportunistic Infection (Infections and infestations) | 18 (19)
Hyperbilirubinemia (Metabolism and nutrition disorders) | 10 (10)
Pain (General disorders) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes